CLINICAL TRIAL: NCT01575847
Title: Adduct Dipstick for Diagnosis of Acetaminophen Toxicity
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other); University of Texas Southwestern Medical Center (Other); Virginia Commonwealth University (Other); Medical University of South Carolina (Other); University of Michigan (Other); University of California, San Francisco (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: Acetaminophen Adduct Dipstick
Record Dates: First submitted 2011-11-23; First posted 2012-04-12 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Acetaminophen Toxicity
Keywords: Acetaminophen; Acetaminophen Toxicity

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Acetaminophen Adduct Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part I: Part 1 will be a feasibility study conducted in the Emergency Department at UAMS and ACH. This Part will test the research use dipsticks and dipstick testing kit in subjects that are having APAP levels obtained as part of their medical evaluation.
  Part 1 20 subjects
  Part I
  Inclusion Criteria:
  Subject is 12-18 years of age. Subject has an APAP level ordered as part of clinical management.
  Exclusion Criteria:
  Previous recent history of APAP overdose in the previous 30 days.
- Part 2: Part 2
  Part 2 will be a non-intervention study in adults presenting to hepatology centers participating in the Acute Liver Failure Study Group (ALFSG). The dipstick will be tested in these subjects and the results will be compared to the HPLC-EC measurement of APAP protein adducts. The results of the dipstick testing will not be used for diagnosis or clinical decision-making.
  Part 2 100 subjects
  Part 2
  Inclusion Criteria:
  Subject is 18 years of age or older. Subject is enrolled in the ALFSG registry.
  Exclusion Criteria:
  None.

SUMMARY:
This study is a non-intervention, clinical study to test "research use only" APAP protein adducts dipsticks in human blood samples. The study will be conducted in two phases. In phase 1, the research use only dipsticks and dipstick testing components will be tested for feasibility in the emergency department at UAMS. Patients will be enrolled that are having an acetaminophen level obtained as part of their medical evaluation. In phase 2, the research use only dipsticks will be tested in centers that participate in the Acute Liver Failure Study Group (ALFSG), a clinical research network funded by the National Institutes of Diabetes, Digestive and Kidney Diseases (NIDDK). Subjects participating in the clinical registry of the ALFSG will be approached for enrollment. These patients all have the diagnosis of acute liver failure or acute liver injury from a variety of etiologies, including APAP. A single blood sample will be obtained and will be aliquoted for 1) testing by the dipstick and 2) testing by high performance liquid chromatography with electrochemical detection (HPLC-EC) analysis for APAP protein adducts. APAP levels will also be determined from the second aliquot of blood. In both Phase 1 and Phase 2, the dipsticks will be read manually and by dipstick readers by independent testers that are not directly involved in the clinical care of the patients. The results of the two dipstick readings will be recorded, will remain confidential and will not be used in the diagnosis or management of the patient. The results of the dipsticks and HPLC-EC assays will be compared to the final patient diagnoses.

ELIGIBILITY:
Part 1

Inclusion Criteria:

* Subject is 12-18 years of age.
* Subject has an APAP level ordered as part of clinical management.

Exclusion Criteria:

* Previous recent history of APAP overdose in the previous 30 days.

Part 2

Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject is enrolled in the ALFSG registry.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Part 1 - Arkansas Children's Hospital ER
  Part 2 - adults presenting to hepatology centers participating in the Acute Liver Failure Study Group (ALFSG).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of dipstick compared to HPLC-EC Method for detecting assays | Each subject will have one sample taken but chart review could last entire hospitalization expected average of 2 weeks
  The primary purpose of this study is to pilot test the study procedures including the dipstick, dipstick instructions, micro-centrifuges, and dipstick readers in a clinical setting and then in the second phase the primary objective will be to compare the results from the dipstick to the currently used method HPLC-EC

CONTACTS AND LOCATIONS:
Overall Officials: Henry Farrar, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences/Arkansas Children's Hospital, Little Rock, Arkansas, United States